CLINICAL TRIAL: NCT03305822
Title: A Study to Evaluate the Pharmacokinetics and Glucodynamics of LY900014 Compared to Humalog Following a Single Dose in Patients With T2DM
Brief Title: A Study of LY900014 in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16640; I8B-MC-ITRU (Other: Eli Lilly and Company); 2017-001305-33 (EudraCT Number)
Record Dates: First submitted 2017-10-05; First posted 2017-10-10 (Actual); Results first posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY900014 (Experimental): Single, subcutaneous (SC) dose of 15 Units (U) LY900014 in one of two study periods
  Interventions: Drug: LY900014
- Insulin Lispro (Humalog) (Active Comparator): Single SC dose of 15 U insulin lispro (Humalog) in one of two study periods
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014
Drug: Insulin Lispro — Administered SC
  Other Names: LY275585; Humalog
  Arms: Insulin Lispro (Humalog)

SUMMARY:
The purpose of this study is to compare LY900014 with insulin lispro (Humalog) in participants with type 2 diabetes mellitus. The study will be conducted in participants with type 2 diabetes on insulin injection therapy to investigate how the body processes LY900014 and the effect of LY900014 on blood sugar levels compared to insulin lispro (Humalog).

Screening is required within 28 days prior to the start of the study. For each participant, the total duration of the clinical trial will be between 3 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female participants with Type 2 Diabetes Mellitus (T2DM) for at least 1 year
* Have a body mass index (BMI) of 18.5 to 35.0 kilogram per meter square (kg/m²)
* Have a glycated hemoglobin (HbA1c) less than (<)9.0 percent (%)
* Have had no episodes of severe hypoglycaemia in the last 6 months

Exclusion Criteria:

* Have a history or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (apart from T2DM), hematological, or neurological disorders capable of significantly altering the absorption, metabolism or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data
* Have a history of renal impairment
* Have a history of deep vein thrombosis of the leg or repeated episodes of deep leg vein thrombosis in first-degree relatives
* Have proliferative retinopathy or maculopathy and/or severe neuropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Neuss, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Leohr J, Dellva MA, Carter K, LaBell E, Linnebjerg H. Ultra Rapid Lispro (URLi) Accelerates Insulin Lispro Absorption and Insulin Action vs Humalog(R) Consistently Across Study Populations: A Pooled Analysis of Pharmacokinetic and Glucodynamic Data. Clin Pharmacokinet. 2021 Nov;60(11):1423-1434. doi: 10.1007/s40262-021-01030-0. Epub 2021 May 27. PMID 34041713
- [Derived] Leohr J, Dellva MA, Coutant DE, LaBell E, Heise T, Andersen G, Zijlstra E, Hermanski L, Nosek L, Linnebjerg H. Pharmacokinetics and Glucodynamics of Ultra Rapid Lispro (URLi) versus Humalog(R) (Lispro) in Patients with Type 2 Diabetes Mellitus: A Phase I Randomised, Crossover Study. Clin Pharmacokinet. 2020 Dec;59(12):1601-1610. doi: 10.1007/s40262-020-00901-2. PMID 32468448

RESULTS

PARTICIPANT FLOW:
Groups:
- LY900014/Humalog: Participants receive a single, subcutaneous (SC) dose of LY900014 with a 3 day washout and a single subcutaneous (SC) 15 U dose of Humalog (insulin lispro)
- Humalog/LY900014: Participants receive a single, subcutaneous (SC) dose of 15 U of Humalog (insulin lispro) with a 3 day washout and a single subcutaneous (SC) LY900014.
Period: Period 1
Arm/Group | LY900014/Humalog | Humalog/LY900014
Started | 20 | 18
Received at Least 1 Dose of Study Drug | 20 | 18
Completed | 20 | 18
Not Completed | 0 | 0
Period: Washout
Arm/Group | LY900014/Humalog | Humalog/LY900014
Started | 20 (Cross-over study. All participants from Period 1 went on to Washout and Period 2.) | 18 (Cross-over study. All participants from Period 1 went on to Washout and Period 2.)
Completed | 20 | 18
Not Completed | 0 | 0
Period: Period 2
Arm/Group | LY900014/Humalog | Humalog/LY900014
Started | 20 | 18
Received at Least 1 Dose of Study Drug | 20 | 18
Completed | 20 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received SC LY900014 or SC Humalog.
Groups:
- Overall: All participants received LY900014 or 15 U Humalog in a crossover design with an approximately 3 day washout period.
Arm/Group | Overall
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 38
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 93.32 (13.03)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under the Plasma Concentration Curve Zero to 10 Hours (AUC[0-10) Following Each Treatment Arm
Description: Pharmacokinetics(PK): Insulin Lispro AUC from zero to 10 hours postdose [AUC(0-10)] following each treatment arm
Time Frame: Predose, 5 minutes (mn), 10mn, 15mn, 20mn, 25mn, 30mn, 35mn, 40mn,45 mn,50mn, 55mn, 60mn, 70mn, 90mn, 120mn, 150mn, 180mn, 240mn, 300mn, 360mn, 420mn, 480mn, 540mn, and 600 minutes(10 hours) postdose
Population: All participants who received at least 1 dose of study drug and have measurable insulin lispro concentrations. No statistical analysis was done, per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour times picomol per liter (pmol*h/L)
Groups:
- LY900014: Participants receive a single, subcutaneous (SC) dose of 15 U LY900014.
- Humalog: Participants receive a single, subcutaneous (SC) dose of 15 U of Humalog (insulin lispro).
Arm/Group | LY900014 | Humalog
Number analyzed (Participants) | 38 | 38
hour times picomol per liter (pmol*h/L) | 1380 (22) | 1280 (24)

2. Secondary Outcome: Pharmacodynamics (PD): Total Amount of Glucose Infused (Gtot) Over Duration of Clamp for Each Treatment Arm
Description: Glucodynamics: Gtot is the total glucose infusion over the clamp duration (10 hours) and is used to measure the study drug action over time as measured by the euglycemic clamp procedure.
Time Frame: Predose, every minute starting from run-in and throughout the duration of the 10 hours
Population: All participants who received at least 1 dose of study drug and had evaluable data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram/kilogram (mg/kg)
Arm/Group | LY900014 | Humalog
Number analyzed (Participants) | 37 | 38
milligram/kilogram (mg/kg) | 749 (59) | 647 (70)

ADVERSE EVENTS:
Time Frame: Baseline until the end of study (60 days)
Groups:
- 15 U LY900014: Participants received a single, subcutaneous (SC) dose 15U LY900014.
- Humalog: Participants received a single, subcutaneous (SC) dose 15 U of Humalog (insulin lispro).
Arm/Group | 15 U LY900014 | Humalog
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/38
Other Adverse Events (participants affected / at risk) | 4/38 | 2/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 U LY900014 (N=38) | Humalog (N=38)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 U LY900014 (N=38) | Humalog (N=38)
Vessel puncture site thrombosis (General disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT03305822/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT03305822/SAP_001.pdf